CLINICAL TRIAL: NCT06934928
Title: Assessing the Efficacy of Repeat, Monthly Treatments of Alexandrite Laser for NF1 Associated Cutaneous Neurofibromas (cNFs)
Brief Title: Assessing the Efficacy of Repeat, Monthly Treatments of Alexandrite Laser for NF1-associated Cutaneous Neurofibromas (cNFs)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Director, Wellman Center for Photomedicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025P000283
Record Dates: First submitted 2025-03-31; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Neurofibromatosis 1 (NF1); Neurofibromatosis Type I
Keywords: Neurofibromatosis; NF1; Cutaneous Neurofibroma; cNF; GentleMax Pro
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatoses | interventions — Lasers, Solid-State; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treated cutaneous neurofibromas (cNFs) (Active Comparator): Participants will receive treatment with laser at a wavelength of 755 nm to the cutaneous Neurofibromas lesion.
  Interventions: Device: GentleMax Pro (with skin cooling); Device: GentleMax Pro (without skin cooling)
- Control cutaneous neurofibromas (cNFs) (No Intervention): A complementary region of cNFs of similar characteristics to the treatment area in the same body region will be selected to serve as an untreated control group.

INTERVENTIONS:
Device: GentleMax Pro (with skin cooling) — Treatment will be performed with the GentleMax Pro laser (755 nm wavelength), which targets hemoglobin.
  A negative pressure hand piece provides temporary, mild suction (~1/2 atm) before laser exposure.
  A pulse fluence of 60-100 J/cm2 (single or double pulse) will be used with 8 mm diameter exposure spot size, and 3 ms pulse duration.
  The laser system includes a dynamic cryogen spray cooling device (DCD) for epidermal protection. A spurt of cryogen cools the epidermis just before arrival of the treatment laser pulse.
  Other Names: Alexandrite Laser; 755 nm Laser; Dynamic Cryogen Spray Cooling Device; DCD
  Arms: Treated cutaneous neurofibromas (cNFs)
Device: GentleMax Pro (without skin cooling) — Treatment will be performed with the GentleMax Pro laser (755 nm wavelength), which targets hemoglobin.
  A negative pressure hand piece provides temporary, mild suction (~1/2 atm) before laser exposure.
  A pulse fluence of 60-100 J/cm2 (single or double pulse) will be used with 8 mm diameter exposure spot size, and 3 ms pulse duration.
  Other Names: Alexandrite Laser; 755 nm Laser
  Arms: Treated cutaneous neurofibromas (cNFs)

SUMMARY:
The goal of this clinical trial is to evaluate the tolerability and effectiveness of multiple treatments of Alexandrite (755 nm) Laser in those with Neurofibromatosis Type 1 (NF1) Cutaneous Neurofibromas (cNFs). The main questions it aims to answer are:

Will performing up to 6 months of treatment sessions with alexandrite laser will result in tolerable local skin reactions and reduction in both individual cNF size by >50% as well as improved cNF appearance in the treated field? If there is a comparison group: Researchers will compare laser treatment with cooling to both laser treatment without cooling and an untreated control see if laser treatments are effective and if cooling makes treatment more tolerable.

Participants will:

* Receive up to 6 monthly laser treatments.
* Complete surveys asking about pain during and after treatments.
* Complete surveys asking about satisfaction with the treatments.
* Undergo 2D photography and 3D imaging of treatment areas.
* Optionally, receive biopsies of up to 6 treated lesions to investigate characteristics of tumors that respond well to treatment as well as non-respondent tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participant is an adult ≥18 years of age.
* Participant has a diagnosis of NF1 based on germline genetic testing or by meeting ≥ 2 the following criteria:
* Family history of NF1
* Six or more light brown ("cafe-au-lait") spots on the skin
* Presence of two or more neurofibromas of any type, or one or more plexiform neurofibromas
* Freckling under the arms or in the groin area
* Two or more pigmented, benign bumps on the eye's iris (Lisch nodules)
* A distinctive bony lesion: dysplasia (abnormal growth) of the sphenoid bone behind the eye, or dysplasia of long bones, often in the lower leg
* Tumor on the optic nerve that may interfere with vision
* Participant is seeking treatment for cNF.
* Participants must have ≥ 12 paired cNF (6 to be treated without DCD, 6 to be treated with DCD) that are visible and measure at least 2 mm in size in the target treatment area. The target treatment area must be amenable to both laser treatments and surveillance with digital and 3D photography. Preferred locations are trunk (back or chest), arms and legs.
* Participant is able and willing to comply with all visit, treatment, and evaluation schedules and requirements.
* Participant is able to understand and provide written informed consent.
* Participant has no concurrent injury or wound in the target area.

Exclusion Criteria:

* Participant cannot give informed consent or adhere to study schedule.
* Participant is Fitzpatrick skin type V-VI.
* Participant is actively tanning during the course of the study.
* For female participants: participant is pregnant.
* Participant has any condition which, in the Investigator's opinion, would make it unsafe (for the participant or study personnel) to treat the participant as part of this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Anytime between initiation of treatment and study completion.
  Treatment will be considered tolerable if <40% of participants treated have a >Grade 2 CTCAE v5 adverse event (AE).

SECONDARY OUTCOMES:
Patient Global Assessment of cNF Improvement (Likert Scale) | Baseline, Day 90, and 30 days after final treatment (up to Day 240).
  Patient rates degree of change of treated cNFs on a scale from -3 (very much worse) to 3 (very large improvement).
Clinician Global Assessment of cNF Improvement (Likert Scale) | Baseline, Day 90, and 30 days after final treatment (up to Day 240).
  Clinician rates degree of change of treated cNFs on a scale from -3 (very much worse) to 3 (very large improvement).
VAS Pain Scale | Baseline, every 30 days (up to Day 240).
  Participants will be asked to rate their pain using a visual analog scale (0 to 10) at each treatment visit and 1 week after each treatment.
Patient Satisfaction | Baseline, Day 90, and 30 days after final treatment (up to Day 240).
  Satisfaction with each treatment modality is rated from 1 (very unsatisfied) to 5 (very satisfied).
Rate of Healing | Baseline, every 30 days (up to Day 240).
  Measured clinically via photography completed by a member of the study team at baseline, and all in-person visits.
cNF Appearance (Height) | Baseline, Day 90, and 30 days after final treatment (up to Day 240).
  Clinically completed 3D Cherry Imaging. Change from baseline in height of cNFs.
cNF Appearance (Volume) | Baseline, Day 90, and 30 days after final treatment (up to Day 240).
  Clinically completed 3D Cherry Imaging. Change from baseline in volume of cNFs.

OTHER OUTCOMES:
Biologic Effect/Histology | 3 months after final treatment session.
  A subset of 2-6 cNFs from the treatment region will be assessed after the final treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. Anderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Wellman Center for Photomedicine, Massachusetts General Hospital, Boston, Massachusetts, United States